CLINICAL TRIAL: NCT06619171
Title: Suicidal Distress in Adolescents With Chronic Pain: Who is at Risk, When, and Why?
Brief Title: Distress in Adolescents With Chronic Pain: Who is at Risk, When, and Why
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Versus Arthritis (Other); Medical Research Foundation (Other); Royal United Hospitals Bath NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PID 17920; IRAS 341501 (Other: Integrated Research Application System (IRAS)); CPMS 64178 (Other: NIHR Central Portfolio Management System (CPMS)); MRF-FEL-CAMPCF-23-105 (Other: Medical Research Foundation & Versus Arthritis)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain
Keywords: Adolescents; Chronic Pain; Distress; Self-Harm; Suicidality; Experience Sampling
MeSH Terms: conditions — Chronic Pain; Self-Injurious Behavior; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Living with chronic pain can be tough for any young person. But while some young people may experience distressing thoughts, others may not. No young person should face these problems alone. So, it's important to better understand who might be more vulnerable to distress, when, and why. That way, healthcare professionals can be there for vulnerable youth when they need it most.

In total, 70 young people with chronic pain (aged 12-19 years) will be invited to take part. Over a 30-day period, they will answer a few questions about their pain and feelings five times per day (experience sampling part) and complete three detailed surveys (at the start, in the middle, and at the end).

This will help the investigators better understand how feelings of pain and distress might change over hours, days, and weeks. Plus, it might reveal which psychological and social factors might bring about these changes.

Answering these questions is vital as it will help healthcare professionals make sure vulnerable young people get the right care at the right time.

DETAILED DESCRIPTION:
This study aims to address the following research questions:

* What are the factors (moderators) that determine why some adolescents with chronic pain may experience suicidal distress but not others, and through which mechanisms (mediators) does chronic pain increase such distress over time?

Primary objective:

The investigators will use the repeated survey data (at day 0, 15, and 31):

* To explore the extent to which pain interference (at baseline) is associated with suicidal distress (primarily hopelessness and entrapment, and secondarily suicidal and self-harm thoughts and behaviours), measured repeatedly over time.

Secondary objectives:

The investigators will use the experience sampling data (5x day/30 days: day 1-30) to explore:

* how the relationship between pain interference and suicidal distress unfolds in the patient's daily life.
* the moderators (collected at baseline, survey data) that determine why some young people with chronic pain may experience suicidal distress over time, but not others.
* the mechanisms (experience sampling items) underpinning the potential relationship between pain interference and suicidal distress in the patient's daily life.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give assent (aged 12-15 years) or informed consent (aged 16 years and older) for participation in the study,
* Parent/guardian is willing to give informed consent for participants aged 12-15 years.
* Adolescents aged 12 to 19 years.
* Were accepted for assessment at a tertiary specialist paediatric pain service, indicating by definition that they experience long-standing, treatment-resistant chronic pain that is functionally interfering.
* Able to read and converse fluently in English.
* Participant is willing to install the m-Path app on a smartphone that runs on Android or iOS to complete the daily assessments. (Please note that a recent Ofcom report has shown that by the age of 12 years, 98% of young people in the UK have their own mobile phone, used by 93% to access social media apps or sites. This supports the nearly universal access of smartphones in this age group)

Exclusion Criteria:

* If some serious acute pathology (e.g., infection, fracture, disease process (e.g., cancer with a potentially fatal trajectory)) or surgical procedure is the cause of the resulting pain complaint.
* If the patient is too psychologically unstable to safely participate in this research, based on clinical judgment (e.g., experiences of acute psychosis)

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We aim to recruit 70 adolescents (aged 12-19 years) with chronic pain.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Hopelessness | day 0 (baseline), 15 (interim survey), and day 31 (final survey)
  Hopelessness Scale for Children (HSC; 17 items) Response options: 1=True, 0=False (total score range: 0-17) The higher the score, the greater the hopelessness for the future.
Entrapment | day 0 (baseline), 15 (interim survey), and day 31 (final survey)
  Short Defeat and Entrapment Scale (4 item entrapment subscale) Response options: 0 = not at all, 1 = a little bit, 2 = moderately, 3 = quite a bit, 4 = extremely like me (total score range: 0-16) Higher scores indicate greater feelings of entrapment.
Suicidal and self-harm thoughts and behaviours | day 0 (baseline), 15 (interim survey), and day 31 (final survey)
  10 separate items on the presence/ absence of suicidal and self-harm thoughts and behaviours.

SECONDARY OUTCOMES:
Hopelessness | day 1 to 30
  single item on hopelessness, assessed repeatedly (5x/30 days) via experience sampling (ESM) Response options: 1 (not at all) - 7 (very much). Higher scores indicate greater feelings of hopelessness
Entrapment | day 1 to 30
  single item on entrapment, assessed repeatedly (5x/30 days) via experience sampling (ESM).
  Response options: 1 (not at all) - 7 (very much). Higher scores indicate greater feelings of entrapment.
Suicidal and self-harm thoughts and behaviours | day 1 to 30
  single items on suicidal and self-harm thoughts and behaviours (5x/30 days), assessed repeatedly via experience sampling (ESM)

CONTACTS AND LOCATIONS:
Overall Officials: Verena Hinze, DPhil, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Bath Centre for Pain Services [BCPS], Bath
  - Oxford Centre for Children and Young People in Pain [OxCYPP], Oxford

IPD SHARING:
Plan to Share IPD: Undecided
A fully de-identified version of the final dataset may be shared with third parties to support future research where it is in the public interest. We will also consider sharing study materials (including codebooks, measures, and analysis code files) openly upon completion of this study.